CLINICAL TRIAL: NCT05325060
Title: Randmised Controlled Trial Comparing Electromagnetically Navigated Versus Conventional Mechanically Aligned Total Knee Arthroplasty
Brief Title: Navigated Versus Convention Total Knee Arthroplasty
Acronym: iNAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RN07OR001
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Arthroplasty, Replacement, Knee; Surgery, Computer-Assisted

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Electromagentically navigated Total knee arthroplasty (Experimental): Patients underwent total knee arthroplasty using the iNav portable EM navigation system (Zimmer GmbH, Winterthur, Switzerland and Medtronic, Minneapolis, MN, USA). The system employs small reference frames attached to the femur and tibia which are incorporated within the primary surgical incision. A standard process of joint registration maps the surface anatomy of the joint. Alignment targets were similar in both groups with a neutral Hip-Knee-Ankle-Axis and the aim to implant both femur and tibial components perpendicular to this in the coronal plane.
  All patients received a cemented posterior stabilized NexGen LPS Flex TKA (Zimmer, Warsaw, Indiana, USA).
  Interventions: Device: Electromagnetically navigated total knee arthroplasty
- Conventional mechanically alligned Total knee arthroplasty (Active Comparator): Participants randomized to the conventional group received a TKA implanted using standard instrumentation.
  All patients received a cemented posterior stabilized NexGen LPS Flex TKA (Zimmer, Warsaw, Indiana, USA).
  Alignment targets were similar in both groups with a neutral Hip-Knee-Ankle-Axis and the aim to implant both femur and tibial components perpendicular to this in the coronal plane.
  Interventions: Device: Conventional total knee arthroplasty

INTERVENTIONS:
Device: Electromagnetically navigated total knee arthroplasty — The navigated group had surgery using the iNav portable EM navigation system (Zimmer GmbH, Winterthur, Switzerland and Medtronic, Minneapolis, MN, USA) and the definitive implant used was NexGen LPS implant (Zimmer Inc, Warsaw, IN, USA), a fixed-bearing bicruciate-sacrificing total condylar implant using traditional instrumentation with no patellar resurfacing
  Arms: Electromagentically navigated Total knee arthroplasty
Device: Conventional total knee arthroplasty — The conventional group received surgery using conventional instrumentation and jigs from the implant manufacturer (Zimmer Inc, Warsaw, IN, USA) and the definitive implant used was NexGen LPS implant (Zimmer Inc, Warsaw, IN, USA), a fixed-bearing bicruciate-sacrificing total condylar implant using traditional instrumentation with no patellar resurfacing
  Arms: Conventional mechanically alligned Total knee arthroplasty

SUMMARY:
The aim of this single blinded randomised control trial study was to assess the accuracy of implantation of components and the clinical outcome and complications with the iNAV electromagnetic navigation system compared with conventional techniques. Secondary outcome measures include Patient reported outcome measures (PROMS) and rates of revision surgery up to 10 years post operatively.

DETAILED DESCRIPTION:
Participants Patients were identified by members of the research team from TKA surgical waiting lists. Patients were invited to participate if they had osteoarthritis of the knee suitable for TKA, were able to provide informed consent, and were aged 18 or over. There were no specific limits imposed on the degree of preoperative coronal or sagittal deformity.

Randomization Overall, 272 patients were screened between July 2007 and August 2010. Of the 272 screened patients, 14 were excluded for other medical reasons, whereas 58 participants decided that they did not want to participate in a research study. The remaining 200 patients were recruited and consented to the study giving a recruitment rate of 74%. Patients were randomized in a 1:1 ratio to either conventional TKA or navigated TKA using a web based computer-generated random number table. Randomization was based on the order of their recruitment and stratified by surgeons to prevent surgeon bias and ensure that similar numbers of patients in each groups were allocated to each surgeon. Randomization was successful in assigning equal preoperative patient demographics between the groups.

Ethical Approval The study was approved by the Glasgow Royal Infirmary Local Ethics Committee and the University of Strathclyde Ethics Committee (07/S0704/6) and approved by the NHS GGC R&D department before commencement of the study.

Surgical Procedure All patients received a cemented posterior stabilized NexGen LPS Flex (Zimmer, Warsaw, Indiana, USA). Participants randomized to the conventional group received a TKA implanted using standard instrumentation, whereas those randomized to the navigated group had surgery using the iNav portable EM navigation system (Zimmer GmbH, Winterthur, Switzerland and Medtronic, Minneapolis, MN, USA). The iNav EM system is imageless and uses small reference frames attached to the femur and tibia which are readily incorporated in the primary incision. There is then a process of joint registration which maps the surface anatomy of the joint. All surgeries including joint surface registration were carried out by, or under the direct supervision of, one of two knee arthroplasty surgeons. Alignment targets were similar in both groups with a neutral HKAA and the aim to implant both femur and tibial components perpendicular to this in the coronal plane.

Ligament balancing was carried out using clinical assessment during the surgical procedure in both groups. In the navigated group, additional information was provided by the system with real-time feedback of the gap in mm between the femoral and tibial component and of the overall HKAA during varus and valgus stress.

Primary outcome measurement Post-operative CT scans were used to determine the accuracy of implantation. CT scan analysis was conducted using Mimics 12.0 software (Materialise, Leuven, Belgium). Measurements of the femoral and tibial component position in the coronal (varus/valgus), sagittal (flexion/extension) and axial (rotational) planes were made. The overall mechanical alignment was also calculated from the addition of the femoral and tibial coronal angles. The combined component rotation was calculated from the addition of the femoral and tibial rotation angles. The rotations were measured using the methods detailed in Berger et al (1998). In the coronal plane the investigators aimed to position both femoral and tibial implants at 90° to the mechanical axis. In the sagittal plane the investigators aimed to position the femoral component with a 5° slope relative to the mechanical axis, in line with the anterior cortex of the distal femur. The tibial component was aimed to be positioned at a 7° slope, as per the manufacturer's guidelines. For femoral rotation the investigators aimed to implant the femoral component in line with the surgical trans-epicondylar axis of the femur. The reference for tibial rotation was a line from the geometric center of the tibia to the center of the tuberosity. Rotational measurements were calculated from a perpendicular line drawn from the posterior surface of the implant. As the tuberosity is 18° externally rotated, the investigators considered an 18° internal rotation of the implant to be a neutral position. (No obvious deformities of the tibia or previous fractures were noted in the study cohort that could have influenced this value.) The investigators considered the desired mechanical axis alignment to be 0° with a range of ± 3°.

Patient-Reported Outcome Measures and Revisions Participants were followed up for 10 years after surgery, with clinical assessments by a blinded independent assessor; range of motion (ROM) was determined using a hand-held goniometer, and knee-specific outcome measures included the American Knee Society Score (AKSS) and Oxford Knee Scores (OKS) and the SF 36 score used as a general health measure (both physical and mental). Revision surgery was also assessed by analyzing the Scottish National Picture Archiving and Communication System. This image archiving system stores all imaging for patients undertaken in the National Health Service (NHS) in Scotland since 2008. It acts as a valuable resource for identifying patients lost to follow-up who have undergone revision surgery in other NHS hospitals in Scotland which may have not been identified.

Statistics A power calculation was performed based in data provided by a randomized controlled trial using infra red optical tracking systems. Bathis et al reported 96% of patients with mechanical leg alignment within 3° of neutral using navigation compared to just 78% with conventional instrumentation . In order to detect a difference of this magnitude with a power of 90% at alpha = 0.05, the investigators would require 82 patients per group, 164 in total. As the primary outcome measure was based on post-operative CT scan the investigators anticipated a higher than average loss to follow-up for the primary outcome measure. The investigators therefore allowed an additional 25% for loss to follow-up, giving a total of 103 patients in each group.

Statistical analysis was performed using SigmaPlot 11.0 (Systat Software Inc). To evaluate differences between the surgical groups either a two sample t test (normally distributed data) or a Mann Whitney test (non parametric data) was performed. A Chi Squared test was used to analysis the male: female ratio. A P value of less that 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* Subjects must be at least 18 years of age and there will be no maximum age limit. The subjects age must be considered suitable by the Investigator for a knee arthroplasty using either of the two systems available in the evaluation.
* Subjects, who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
* Subjects, who, in the opinion of the investigator, are able to understand this investigation, co-operate with the investigation procedures and are willing to return to the hopsital for all the required post-operative follow-ups.
* Subjects who require a knee arthroplasty for primary surgical management of the idiopathic osteoarthritis.
* Subjects, who in the opinion of the Investigator, are considered to be suitable for treatment with a NexGen LPS Flex Total Knee Replacement.

Exclusion Criteria:

* Subjects who, in the opinion of the investigator, have an existing condition that would compromise their participation and follow-up in the study
* Subjects who require revision total knee arthroplasty surgery
* Subjects with any tibial deformity requiring tibial component augmentation.
* Subjects whom, in the opinion of the Investigator, require a constratined prosthesis.
* Subjects with inflammatory polyarthritis.
* Subjects with disorders of the feet, ankles, hips, or spine caising significant abnormal gait or significant pain.
* Subjects with osteoarthritis of the contralateral knee causing significant abnormal gait or significant pain.
* Subjects with poorly functioning contralateral total knee replacement causing significant abnormal gait or significant pain. Subjects with a well functioning contralateral total knee replacement will not be excluded.
* Subjects with neurological conditions affecting movement.
* Subjects with a pathology which, in the opinion of the Investigator, will adversely affect healing.
* Subjects with other disorders which, in the opinion of the Investigator, will/could impair rehabilitation.
* Contra-indications for the use of the device, as detailed in the package insert.
* Women who are pregnant
* Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes.
* Subjects who are currently invovled in another clinical study with an investigational product.
* Subjects who are currently invovled in any injury litigation claims.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-06-25 (Actual); Primary Completion 2010-12-07 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Knee coronal plane allignment | 3 months post operatively
  The primary outcome measure for this study was alignment within 3 degrees of neutral mechanical alignment at three months after surgery

SECONDARY OUTCOMES:
Oxford knee score | Up to 10 years post operatively
  Patient reported outcome measure validated for total knee arthroplasty
American Knee Society Score | Up to 10 years post operatively
  Patient reported outcome measure validated for total knee arthroplasty
Short Form 36 Health Survey Questionnaire (SF-36) | Up to 10 years post operatively
  Validated self reported outcome measure of health
Range of motion | 10 years post operatively
  Measured by research assistant post operatively using established techniques
All cause revision surgery | 10 years post operatively
  Examines re-intervention rates for any cause post-operatively. We defined revision using the United Kingdom National Joint registery definition of any intervention that results in the addition, removal or exchange of any component of the primary implant

CONTACTS AND LOCATIONS:
Overall Officials: Mark JG Blyth, Mr, Principal Investigator — NHS Greater Glasgow and Clyde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Decking R, Markmann Y, Fuchs J, Puhl W, Scharf HP. Leg axis after computer-navigated total knee arthroplasty: a prospective randomized trial comparing computer-navigated and manual implantation. J Arthroplasty. 2005 Apr;20(3):282-8. doi: 10.1016/j.arth.2004.09.047. PMID 15809943
- [Background] Chin PL, Yang KY, Yeo SJ, Lo NN. Randomized control trial comparing radiographic total knee arthroplasty implant placement using computer navigation versus conventional technique. J Arthroplasty. 2005 Aug;20(5):618-26. doi: 10.1016/j.arth.2005.04.004. PMID 16309998
- [Background] Haaker RG, Stockheim M, Kamp M, Proff G, Breitenfelder J, Ottersbach A. Computer-assisted navigation increases precision of component placement in total knee arthroplasty. Clin Orthop Relat Res. 2005 Apr;(433):152-9. doi: 10.1097/01.blo.0000150564.31880.c4. PMID 15805951
- [Background] Bolognesi M, Hofmann A. Computer navigation versus standard instrumentation for TKA: a single-surgeon experience. Clin Orthop Relat Res. 2005 Nov;440:162-9. doi: 10.1097/01.blo.0000186561.70566.95. PMID 16239801
- [Background] Bathis H, Perlick L, Tingart M, Luring C, Zurakowski D, Grifka J. Alignment in total knee arthroplasty. A comparison of computer-assisted surgery with the conventional technique. J Bone Joint Surg Br. 2004 Jul;86(5):682-7. doi: 10.1302/0301-620x.86b5.14927. PMID 15274263
- [Result] Clark AN, Hounat A, O'Donnell S, May P, Doonan J, Rowe P, Jones BG, Blyth MJG. Electromagnetic Navigated Versus Conventional Total Knee Arthroplasty-A Five-Year Follow-Up of a Single-Blind Randomized Control Trial. J Arthroplasty. 2021 Oct;36(10):3451-3455. doi: 10.1016/j.arth.2021.06.007. Epub 2021 Jun 12. PMID 34226082
- [Result] Blyth MJ, Smith JR, Anthony IC, Strict NE, Rowe PJ, Jones BG. Electromagnetic navigation in total knee arthroplasty-a single center, randomized, single-blind study comparing the results with conventional techniques. J Arthroplasty. 2015 Feb;30(2):199-205. doi: 10.1016/j.arth.2014.09.008. Epub 2014 Sep 16. PMID 25263246
- [Result] Smith JR, Rowe PJ, Blyth M, Jones B. The effect of electromagnetic navigation in total knee arthroplasty on knee kinematics during functional activities using flexible electrogoniometry. Clin Biomech (Bristol). 2013 Jan;28(1):23-8. doi: 10.1016/j.clinbiomech.2012.09.006. Epub 2012 Oct 18. PMID 23083704